CLINICAL TRIAL: NCT04080635
Title: Evaluation of the Predictive Value of Early Serum Trough Concentrations and Anti-drug Antibodies of Brodalumab and the Development of Concentration-response Curve of Brodalumab of Psoriasis Patients.
Brief Title: Therapeutic Drug Monitoring of Brodalumab in Psoriasis Patients (BIOLOPTIM-BRO)
Acronym: BIOLOPTIM-BRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-03913 - BIOLOPTIM-BRO
Record Dates: First submitted 2019-07-19; First posted 2019-09-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis; Therapeutic drug monitoring; Brodalumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: A prospective, open label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care - brodalumab (Experimental): Patients will continue to receive brodalumab according to standard care dosing regimen, i.e. loading dose first (210mg), once a week for 2 weeks (210mg), then a regular dose regimen (210mg) every 2 weeks.
  Interventions: Procedure: Venapuncture; Other: Patient questionnaires

INTERVENTIONS:
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of brodalumab
Other: Patient questionnaires — The study participant will complete the Dermatology Quality of Life Index (DLQI) and EQ5D5L

SUMMARY:
Biologics, such as brodalumab, are currently the most effective treatment option for patients with moderate-to-severe psoriasis. But they are costly for health care systems and prescribed according to a 'one dose fits all' dosing regimen, leading to potential over- and undertreatment. Within this study we aim to investigate the predictive value of early serum trough levels of brodalumab and determine the therapeutic window of brodalumab in psoriasis patients.

DETAILED DESCRIPTION:
Patients will be included after siging informed consent. After inclusion, patients will continue on standard dosing schedule of brodalumab (i.e. one loading dose first (210mg), once a week for 2 weeks (210mg), then a regular dose regimen (210mg) every 2 weeks). During each study visit, blood will be taken in order to quantify Ctroughs and/or anti-drug antibodies towards brodalumab. In addition, the Psoriasis Severity and Area Index (PASI) and the Investigator's Global Assessment (IGA) score will be evaluated by a physician. Patients complete the Dermatology Life Quality Index (DLQI) and European quality of life EQ-5D instrument at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a clinical or histological diagnosis of chronic plaque-type psoriasis
2. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

1. Participants who have currently a predominant nonplaque form of psoriasis
2. Participants who are pregnant, nursing or planning a pregnancy
3. Participants who are unable or unwilling to undergo multiple venapunctures
4. Participants who are treated according to a different dosing schedule than standard dosing of brodalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of early serum trough concentrations of brodalumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 25 based on serum trough concentrations measurements taken from week 0, 1, 2, 3 and/or 4.
Predictive value of early anti-drug antibodies of brodalumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 24 based on anti-drug antibodies measurements taken from week 0, 1, 2, 3 and/or 4.
The development of a therapeutic window of brodalumab in psoriasis | Week 0 until week 52 of treatment
  Defining a therapeutic window for brodalumab based on serum trough levels corresponding with adequate clinical response.

SECONDARY OUTCOMES:
DLQI | Week 0 until week 52 of treatment
  The DLQI (Dermatology Life Quality Index) (range 0-30) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the disease on participant's QoL. It is a ten item questionnaire that, in addition to evaluated overall QoL, can be used to assess six different aspects that may affect QoL: 1) symptoms and feelings, 2) daily activities, 3) leasure, 4) work or school performances, 5) personal relationships, and 6) treatment.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
EQ5D5L | Week 0 until week 52 of treatment
  EQ5DL comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EQ VAS | Week 0 until week 52 of treatment
  The EQ VAS (Visual Analogue Scale) (range 0-10) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Ghent
Locations (7):
- Belgium (7):
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - AZ Sint-Lucas, Ghent, Oost-Vlaanderen
  - University Hospital of Ghent, Ghent, Oost-Vlaanderen
  - Private Practice Dermatology, Maldegem, Oost-Vlaanderen
  - University Hospital, Leuven, Vlaams-Brabant
  - AZ Sint-Jan, Bruges, West-Vlaanderen
  - AZ Delta Rembert, Torhout, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No